CLINICAL TRIAL: NCT04937699
Title: Efficacy and Safety of Sequential Monotherapy of Ticagrelor and Clopidogrel in Patients Undergoing Percutaneous Coronary Intervention With Acute Coronary Syndrome
Brief Title: Sequential MonotherApy of TicagrElor and Clopidogrel After Coronary Intervention
Acronym: MATE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-MATE-01
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: ticagrelor; monotherapy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-DAPT of Ticagrelor plus aspirin (DAPT) (Active Comparator): Patients will receive Standard-DAPT of Ticagrelor plus aspirin for 1month after PCI and continue to receive standard-DAPT till 1 year in this arm after as followed:
  Ticagrelor 90mg bid+Aspirin 100mg qd for 1month; Ticagrelor 90mg bid+Aspirin 100mg qd for another 11 months;
  Interventions: Drug: Standard-DAPT of Ticagrelor plus aspirin
- Sequential monotherapy of Ticagrelor and Clopidogrel (SAPT) (Experimental): Patients will receive Standard-DAPT of Ticagrelor plus aspirin for 1month after PCI and switch to ticagrelor monotherapy in the following 5 months, and then further de-escalated to clopidogrel monotherapy till 1 year in this arm as followed:
  Ticagrelor 90mg bid+Aspirin 100mg qd for 1 month; Ticagrelor 90mg bid, for 5 months; clopidogrel 75mg qd, for 6 months.
  Interventions: Drug: Sequential monotherapy of Ticagrelor and clopidogrel

INTERVENTIONS:
Drug: Standard-DAPT of Ticagrelor plus aspirin — Ticagrelor 90mg bid+Aspirin 100mg qd for 1 month after PCI, Randomized subjects continue for another 11 months
  Other Names: DAPT
  Arms: Standard-DAPT of Ticagrelor plus aspirin (DAPT)
Drug: Sequential monotherapy of Ticagrelor and clopidogrel — Ticagrelor 90mg bid+Aspirin 100mg qd for 1 month after PCI, Randomized subjects switch to ticagrelor 90mg bid for 5 months; then clopidogrel 75mg qd, for another 6 months.
  Other Names: SAPT
  Arms: Sequential monotherapy of Ticagrelor and Clopidogrel (SAPT)

SUMMARY:
The MATE study is a randomized, multicenter, open-label, investigator-initiated clinical trial aimed to evaluate efficacy and safety of sequential monotherapy of ticagrelor and clopidogrel in patients with acute coronary syndrome (ACS) after coronary intervention. Standard DAPT of aspirin plus ticagrelor will be given for the first 1 month after PCI. After 1 month, event-free subjects will be randomized at 1:1 ratio into receiving standard DAPT (DAPT) until 12months , or switch to ticagrelor monotherapy for another 5 months , and further de-escalated to monotherapy of clopidogrel for the last 6 months(SAPT).

DETAILED DESCRIPTION:
Compared with clopidogrel, ticagrelor inhibit platelet aggregation faster and stronger, and significantly reduce the risk of cardiovascular and cerebrovascular adverse events. In recent years, it has been given the strongest recommendation for antiplatelet therapy in ACS patients. Nevertheless, it was shown that excessive bleeding events significantly affect its antithrombotic advantage and better safety by downgrading regimen can seek more net clinical benefit. However, there are still huge controversies regarding the degree or timing of the downgrading regimen.

GLOBAL LEADERS study shortened the course of DAPT after PCI to 1 month in "all-comer" population of coronary heart disease , and then downgraded to ticagrelor monotherapy and continued 23 months. At 12 months, compared with standard DAPT, there was neither increased risk of thrombotic events, nor significant reduction in BARC3 or type 5 major bleeding events, which suggested satisfactory safety of 1-month DAPT, and relative insufficiency de-escalation. The most recent STOPDAPT-2 ACS study not only adapted 1-month DAPT (prasugrel or clopidogrel + aspirin) in ACS patients, but also directly downgraded to clopidogrel monotherapy. Compared with standard DAPT of clopidogrel + aspirin, clopidogrel monotherapy significantly reduces the risk of bleeding, however, it also increases the thrombotic risk. Overrall, the investigators believe that de-escalated antiplatelet therapy are most suitable in ACS patients undergoing PCI. Short-course DAPT based on potent P2Y12 inhibitors will not increase the thrombotic risk, but continuous application of one single P2Y12 receptor antagonists may be difficult to take into account both the antithrombotic efficacy and bleeding benefit, while the sequential monotherapy of ticagrelor and clopidogrel may be more conducive to balancing the two needs.

In summary, the current project aimed at"all-comer"population of ACS, for the first time proposed a de-escalated antiplatelet regimen of sequential monotherapy of ticagrelor and clopidogrel. In this project, ticagrelor monotherapy will be used 1 month after PCI, and the anti-platelet strength will be further downgraded 5 months later to clopidogrel (75 mg) monotherapy till 1 year, which is supposed to achieve a better safety benefit and a non-inferior efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Acute coronary syndrome was diagnosed upon admission;
3. Administered ticagrelor for at least 30 days after successful PCI with implantation of a current-generation drug-eluting stent(s)
4. Agree to the study protocol and the schedule of clinical follow-up, and provides informed, written consent

Exclusion Criteria:

1. Implanted with first-generation DES or bioabsorbable stent(s) during hospitalization;
2. Patients with active pathological bleeding (such as peptic ulcer or intracranial hemorrhage);
3. History of intracranial hemorrhage, intracranial neoplasms, intracranial vascular malformations or hemangioma
4. High potential risk of major bleeding, such as acute or chronic gastrointestinal ulcers or other gastrointestinal diseases, alignant tumors, etc.;
5. Thrombolytic therapy within 24 hours of index PCI;
6. Planned coronary revascularization (surgical or percutaneous) within 30 days;
7. Allergic to ticagrelor, clopidogrel or aspirin and any excipients;
8. Inability to tolerate 12-month DAPT (ticagrelor+aspirin) for any reason;
9. Cardiogenic shock or hemodynamic instability;
10. Diagnosed as active hepatitis or liver cirrhosis upon admission;
11. Suffer from a known serious progressive disease (e.g. progressive cancer, chronic obstructive lung disease, etc.;) or estimated survival time<12 months ;
12. Platelet count<100000 /mm3;
13. Dialysis-dependent renal failure；
14. Required use of oral anticoagulation (warfarin or other factor II or factor X inhibitors);
15. Pregnant or plan to be pregnant within 1 year;
16. Any condition that may interfere with any study procedures, such as dementia, immobility, alcohol use, etc;
17. Participating in any other clinical trial of an investigational drug or device that has not met its primary endpoint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2690 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
NACCE | 1-12months after PCI (11 months after randomization)
  Cumulative incidence of cardiovascular death, myocardial infarction, stroke (ischaemic, haemorrhagic, or unknown aetiology), definite stent thrombosis and bleeding type 2, 3 or 5 according to the Bleeding Academic Research Consortium (BARC) criteria.

SECONDARY OUTCOMES:
MACCE | 1-12months after PCI (11 months after randomization)
  The Key secondary endpoint for ischemic outcome is cumulative incidence of cardiovascular death, non-fatal myocardial infarction,definite stent thrombosis or stroke (ischaemic, haemorrhagic, or unknown aetiology)

OTHER OUTCOMES:
BARC types 2,3 or 5 bleeding | 1-12months after PCI (11 months after randomization)
  The Key secondary endpoint for bleeding outcome is cumulative incidence of BARC types 2,3 or 5 bleeding according to the Bleeding Academic Research Consortium (BARC) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sun, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The deidentified data will be shared after publication of first manuscript
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Watanabe H, Morimoto T, Natsuaki M, Yamamoto K, Obayashi Y, Ogita M, Suwa S, Isawa T, Domei T, Yamaji K, Tatsushima S, Watanabe H, Ohya M, Tokuyama H, Tada T, Sakamoto H, Mori H, Suzuki H, Nishikura T, Wakabayashi K, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 ACS Investigators. Comparison of Clopidogrel Monotherapy After 1 to 2 Months of Dual Antiplatelet Therapy With 12 Months of Dual Antiplatelet Therapy in Patients With Acute Coronary Syndrome: The STOPDAPT-2 ACS Randomized Clinical Trial. JAMA Cardiol. 2022 Apr 1;7(4):407-417. doi: 10.1001/jamacardio.2021.5244. PMID 35234821
- [Result] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Result] Wu B, Lin H, Tobe RG, Zhang L, He B. Ticagrelor versus clopidogrel in East-Asian patients with acute coronary syndromes: a meta-analysis of randomized trials. J Comp Eff Res. 2018 Mar;7(3):281-291. doi: 10.2217/cer-2017-0074. Epub 2017 Nov 2. PMID 29094604
- [Result] Wang HY, Li Y, Xu XM, Li J, Han YL. Impact of Baseline Bleeding Risk on Efficacy and Safety of Ticagrelor versus Clopidogrel in Chinese Patients with Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention. Chin Med J (Engl). 2018 Sep 5;131(17):2017-2024. doi: 10.4103/0366-6999.239306. PMID 30127210
- [Result] Li P, Gu Y, Yang Y, Chen L, Liu J, Gao L, Qin Y, Cai Q, Zhao X, Wang Z, Ma L. Low-dose ticagrelor yields an antiplatelet efficacy similar to that of standard-dose ticagrelor in healthy subjects: an open-label randomized controlled trial. Sci Rep. 2016 Aug 24;6:31838. doi: 10.1038/srep31838. PMID 27554803
- [Result] Orme RC, Parker WAE, Thomas MR, Judge HM, Baster K, Sumaya W, Morgan KP, McMellon HC, Richardson JD, Grech ED, Wheeldon NM, Hall IR, Iqbal J, Barmby D, Gunn JP, Storey RF. Study of Two Dose Regimens of Ticagrelor Compared With Clopidogrel in Patients Undergoing Percutaneous Coronary Intervention for Stable Coronary Artery Disease. Circulation. 2018 Sep 25;138(13):1290-1300. doi: 10.1161/CIRCULATIONAHA.118.034790. Epub 2018 Jul 24. PMID 29930021
- [Result] Park DW, Lee PH, Jang S, Lim HS, Kang DY, Lee CH, Ahn JM, Yun SC, Park SW, Park SJ. Effect of Low-Dose Versus Standard-Dose Ticagrelor and Clopidogrel on Platelet Inhibition in Acute Coronary Syndromes. J Am Coll Cardiol. 2018 Apr 10;71(14):1594-1595. doi: 10.1016/j.jacc.2018.02.010. No abstract available. PMID 29622168
- [Result] Levine GN, Jeong YH, Goto S, Anderson JL, Huo Y, Mega JL, Taubert K, Smith SC Jr. Expert consensus document: World Heart Federation expert consensus statement on antiplatelet therapy in East Asian patients with ACS or undergoing PCI. Nat Rev Cardiol. 2014 Oct;11(10):597-606. doi: 10.1038/nrcardio.2014.104. Epub 2014 Aug 26. PMID 25154978
- [Result] Vranckx P, Valgimigli M, Juni P, Hamm C, Steg PG, Heg D, van Es GA, McFadden EP, Onuma Y, van Meijeren C, Chichareon P, Benit E, Mollmann H, Janssens L, Ferrario M, Moschovitis A, Zurakowski A, Dominici M, Van Geuns RJ, Huber K, Slagboom T, Serruys PW, Windecker S; GLOBAL LEADERS Investigators. Ticagrelor plus aspirin for 1 month, followed by ticagrelor monotherapy for 23 months vs aspirin plus clopidogrel or ticagrelor for 12 months, followed by aspirin monotherapy for 12 months after implantation of a drug-eluting stent: a multicentre, open-label, randomised superiority trial. Lancet. 2018 Sep 15;392(10151):940-949. doi: 10.1016/S0140-6736(18)31858-0. Epub 2018 Aug 27. PMID 30166073